CLINICAL TRIAL: NCT03468660
Title: Auditory Temporal Processes, Speech Perception and Aging
Brief Title: Auditory Temporal Processes in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Sandra Gordon Salant, Professor, University of Maryland, College Park
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMDCP
Record Dates: First submitted 2018-03-06; First posted 2018-03-16 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Auditory Perceptual Disorders; Aging Problems
Keywords: Accented speech perception
MeSH Terms: conditions — Auditory Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: Experimental group Active control group Passive control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Auditory training with feedback
  Interventions: Behavioral: Auditory training with feedback
- Passive control group (No Intervention): Pre-post testing only; no training
- Active Control group (Active Comparator): Listening task with no feeback
  Interventions: Behavioral: Listening paradigm with no feedback

INTERVENTIONS:
Behavioral: Auditory training with feedback — Experimental group receives phoneme-level and sentence-level training with feedback
  Arms: Experimental group
Behavioral: Listening paradigm with no feedback — Active controls listen to acoustic stimuli with no feedback
  Arms: Active Control group

SUMMARY:
Older people experience great difficulty understanding speech, especially accented English, and this problem is expected to increase with the influx of immigrants who provide services to the elderly population. The research examines the underlying factors that contribute to older listeners' difficulty understanding accented speech, including those associated with age-related hearing loss, changes in processing in auditory pathways in the brain, and general cognitive decline. The investigation also evaluates the efficacy of training strategies to improve understanding of accented English by older people. Outcomes of this research are expected to improve communication between senior citizens and those with whom they interact daily, and thereby improve quality of life for the older segment of the Nation's population.

DETAILED DESCRIPTION:
This research program in speech perception and auditory psychophysics examines the hypothesis that many of the predominant difficulties in speech understanding of elderly listeners are related to underlying problems in auditory temporal processing. One form of degraded speech that is particularly difficult for elderly listeners to perceive is accented English. Alterations of speech stress and timing with accent may be viewed as a form of degradation in temporal aspects of speech prosody, and this type of temporal distortion is the focus of investigation in the next project period. Moreover, psychoacoustic results demonstrate that large age-related difficulties in temporal processing exist for the perception of auditory tempo and rhythmic characteristics of sequential stimulus patterns featuring a stressed tone. Listener processing difficulty could be attributed to peripheral and/or central processing mechanisms, as well as various cognitive factors, including the degree of familiarity with prosodic features of different native languages. The project examines the relative contribution of peripheral hearing impairment, type of stimulus temporal complexity and cognitive demand, and the linguistic background experience of listeners on the processing of temporal prosody cues in speech and non-speech stimulus patterns. The project associated with this clinical trial examines the efficacy of auditory training paradigms with stimuli that feature temporal contrasts for improving perception of accented English and non-speech sequences by older people. The research described in this application seeks to address one goal outlined by the National Institute on Aging: to develop effective interventions to maintain health and function and prevent or reduce the burden of age-related diseases, disorders, and disabilities. The approach in this research program involves (a) an assessment of the problems encountered in daily activities by the elderly population, (b) an analysis of specific task demands in relation to individual capabilities, and (c) basic research on sensory and perceptual changes with age and on the ameliorating effects of emerging technologies (including rehabilitation). This three-dimensional approach is expected to further progress toward improving communication and health-related quality of life for senior citizens.

ELIGIBILITY:
Inclusion Criteria:

* Age and hearing sensitivity:
* Younger listeners (18-40 years) with normal hearing;
* Older listeners (65-80 years) with normal hearing;
* Older listeners (65-80 years) with bilateral, mild-to-moderate sensorineural hearing loss.
* High School Diploma,
* native speaker of English (based on self-report)
* normal middle-ear function (based on tympanometry)
* normal cognitive function (based on score on Montreal Cognitive Assessment)
* good-to-excellent word recognition scores (based on Northwestern University Test # 6 word recognition scores presented in quiet at suprathreshold levels).

Exclusion Criteria:

* non-native speaker of English,
* motor and/or speech disorders that prevent participant from providing a time-locked response,
* presence of middle ear disease or conductive hearing loss,
* presence of severe or profound hearing loss,
* presence of poor word recognition scores,
* cognitive impairment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Recognition of accented speech stimuli used for training | 1 day
  Scale: Accented words (n = 160) and accented sentences (n = 35 sentences) used in training; construct: measures percent correct recognition; minimum score = 0%, maximum score = 100%. Higher values are considered a better outcome

SECONDARY OUTCOMES:
Generalization of benefit in recognizing accented speech | 1 day
  Scale: Accented words (n = 48) and accented sentences (n = 10 sentences) with new talker and speech stimuli not used in training. Construct measures percent correct recognition score for accented words and sentences not used in training, with minimum = 0% and maximum = 100%. Better performance is a higher percent correct score.
Retention of benefit in recognizing accented speech | through study completion, an average of two weeks
  Scale: Accented words (n = 64) and accented sentences (n = 90). For words: familiar words and familiar talkers (n = 32) and new talkers and new words (n = 32). For sentences: familiar talkers and words (used in training; n = 40), new talkers and new lists not heard before (n = 20), and talkers and sentences heard before but not used in training (n = 30). Construct: percent correct recognition for trained talker and lists, new talkers and new stimuli, and familiar talkers and lists not used in training. Construct: percent correct recognition (min = 0%, max = 100%), with better performance a higher recognition score.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Gordon-Salant, Ph.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon-Salant S, Yeni-Komshian GH, Bieber RE, Jara Ureta DA, Freund MS, Fitzgibbons PJ. Effects of Listener Age and Native Language Experience on Recognition of Accented and Unaccented English Words. J Speech Lang Hear Res. 2019 Apr 26;62(4S):1131-1143. doi: 10.1044/2018_JSLHR-H-ASCC7-18-0122. PMID 31026190
- [Background] Bieber RE, Yeni-Komshian GH, Freund MS, Fitzgibbons PJ, Gordon-Salant S. Effects of listener age and native language on perception of accented and unaccented sentences. J Acoust Soc Am. 2018 Dec;144(6):3191. doi: 10.1121/1.5081711. PMID 30599683
- [Result] Bieber RE, Gordon-Salant S. Adaptation to novel foreign-accented speech and retention of benefit following training: Influence of aging and hearing loss. J Acoust Soc Am. 2017 Apr;141(4):2800. doi: 10.1121/1.4980063. PMID 28464671
- [Result] Fitzgibbons PJ, Gordon-Salant S. Age effects in discrimination of intervals within accented tone sequences differing in accent type and sequence presentation rate. J Acoust Soc Am. 2016 Nov;140(5):3819. doi: 10.1121/1.4967512. PMID 27908085
- [Result] Gordon-Salant S, Yeni-Komshian GH, Pickett EJ, Fitzgibbons PJ. Perception of contrastive bi-syllabic lexical stress in unaccented and accented words by younger and older listeners. J Acoust Soc Am. 2016 Mar;139(3):1132-48. doi: 10.1121/1.4943557. PMID 27036250
- [Result] Gordon-Salant S, Yeni-Komshian GH, Fitzgibbons PJ, Cohen JI. Effects of age and hearing loss on recognition of unaccented and accented multisyllabic words. J Acoust Soc Am. 2015 Feb;137(2):884-97. doi: 10.1121/1.4906270. PMID 25698021
- [Result] Gordon-Salant S, Yeni-Komshian GH, Fitzgibbons PJ, Cohen JI, Waldroup C. Recognition of accented and unaccented speech in different maskers by younger and older listeners. J Acoust Soc Am. 2013 Jul;134(1):618-27. doi: 10.1121/1.4807817. PMID 23862836
- [Result] Gordon-Salant S, Yeni-Komshian GH, Fitzgibbons PJ. Recognition of accented English in quiet and noise by younger and older listeners. J Acoust Soc Am. 2010 Nov;128(5):3152-60. doi: 10.1121/1.3495940. PMID 21110610
- [Result] Gordon-Salant S, Yeni-Komshian GH, Fitzgibbons PJ, Schurman J. Short-term adaptation to accented English by younger and older adults. J Acoust Soc Am. 2010 Oct;128(4):EL200-4. doi: 10.1121/1.3486199. PMID 20968326
- [Result] Gordon-Salant S, Yeni-Komshian GH, Fitzgibbons PJ. Recognition of accented English in quiet by younger normal-hearing listeners and older listeners with normal-hearing and hearing loss. J Acoust Soc Am. 2010 Jul;128(1):444-55. doi: 10.1121/1.3397409. PMID 20649238
- [Result] Fitzgibbons PJ, Gordon-Salant S. Age-related differences in discrimination of temporal intervals in accented tone sequences. Hear Res. 2010 Jun 1;264(1-2):41-7. doi: 10.1016/j.heares.2009.11.008. Epub 2009 Dec 3. PMID 19931608